CLINICAL TRIAL: NCT00305513
Title: Effectiveness of Rehabilitation (Phasic Alerting and Visual Spatial Scanning Training) on the Recovery of Patients Post Right Stroke With Unilateral Spatial Neglect: Using Functional Imaging PET and Standardized Neurobehavioral and Functional Tests
Brief Title: Effectiveness of Rehabilitation on the Recovery of Patients Post Right Stroke With Unilateral Spatial Neglect
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-17.02.06-HMO-CTIL
Record Dates: First submitted 2006-03-21; First posted 2006-03-22 (Estimated); Last update posted 2010-06-03 (Estimated); Status verified 2006-03

CONDITIONS: Cerebrovascular Accident; Perceptual Disorders
Keywords: right hemispheric CVA; neglect; phasic alert treatment; PET scan; patients post right hemispheric CVA (stroke)
MeSH Terms: conditions — Stroke; Perceptual Disorders

INTERVENTIONS:
Procedure: The phasic alerting treatment

SUMMARY:
Unilateral spatial neglect (USN) is believed to be a disorder of attention, characterized by impairment in the ability to perceive or respond to stimuli presented to the contralesional space, and which is not attributable to significant sensory or motor deficits. USN has serious consequences for rehabilitation and long term disabilities. Efforts have been made to clarify both the theoretical basis of this phenomenon and the rehabilitation methods that will be best in improving function. The purpose of this study is to try and contribute to both efforts by examining treatment effectiveness of two methods; one targeting general arousal (phasic alerting), and the other targeting increasing awareness to left side stimuli and habit changes. Functional neuroimaging methods (PET [positron emission tomography] and fMRI [functional magnetic resonance imaging]) have been applied to understand the functional anatomy of the brain during mental processes. Only a few attempts have been made to use functional neuroimaging in patients with neurological deficits such as USN, usually speculations are made based on findings with healthy participants to explain this disorder. This study's aim is to examine the functional reorganization of the attentional network in the brain of USN patients while performing visual tasks, by means of functional neuroimaging techniques, in light of specific rehabilitation techniques.

Patients will be examined before and after 3 weeks of rehabilitation both using standardized neurobehavioral tests and PET imaging procedures.

DETAILED DESCRIPTION:
Procedure:

Inclusion criteria:

* first time right hemispheric stroke (ischemic);
* 2-6 weeks post stroke incident;
* ages 25-85;
* right hand dominance;
* minimum education of 6 years;
* do not suffer from field cut deficit such as hemi-anopsia;
* without other known neurological disorders (e.g., Parkinson's disease, aphasia);
* without severe systemic conditions (e.g., malignancies, AIDS, congestive heart failure, substance abuse);
* did not take additional medications that could affect the central nervous system; without dementia;
* without mental illness;
* the patients or their legal guardians have to give informed consent.

Participants:

* six patients will be recruited and randomly allocated to one of the treatment groups (phasic alerting or standard visual spatial training treatment provided in the OT department).

Patients will undergo thorough evaluation of neglect and will undergo PET procedure before being transferred to rehabilitation. Patient will receive intensive rehabilitation for 15 sessions of the cognitive treatment and 15 session of motor training. After this period patient will undergo another PET procedure to assess any changes in brain activation. Patient will then return to rehabilitation as needed.

ELIGIBILITY:
Inclusion Criteria:

* First time right hemispheric stroke (ischemic)
* 2 - 6 weeks post stroke incident
* Ages 25 - 85
* Right hand dominance
* Minimum education of 6 years
* The patients or their legal guardians have to give informed consent
* Does not suffer from field cut deficit such as hemi-anopsia
* Without other known neurological disorders (e.g., Parkinson's disease, aphasia)
* Without severe systemic conditions (e.g., malignancies, AIDS, congestive heart failure, substance abuse)
* Does not take additional medications that could affect the central nervous system
* Without dementia
* Without mental illness

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)

PRIMARY OUTCOMES:
This study's aim is to examine the functional reorganization of the attentional network in the brain of USN patients while performing visual tasks, by means of functional neuroimaging techniques, in light of specific rehabilitation techniques.

SECONDARY OUTCOMES:
The aim of this study is to try and contribute to both efforts by examining treatment effectiveness of two methods; one targeting general arousal (phasic alerting), and the other targeting increasing awareness to left side stimuli and habit changes.

CONTACTS AND LOCATIONS:
Overall Officials: Zeev Meiner, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel